CLINICAL TRIAL: NCT04893005
Title: Knowledge Level of Pelvic Floor in Different Age Groups
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: pelvic floor
Record Dates: First submitted 2021-05-16; First posted 2021-05-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor,; knowledge,; Turkey
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Having knowledge and awareness about pelvic floor muscles and pelvic floor dysfunctions makes it easier for individuals to understand their own body and the treatment provided to them by healthcare professionals (Fante, 2019). In the literature, there are studies investigating the knowledge and awareness levels of different participant groups about pelvic floor and pelvic floor dysfunctions (Parden, 2016; Hill, 2017; Falvey, 2020). It has been shown that most women lack knowledge of pelvic floor muscle dysfunction, do not understand treatment options for the pelvic floor, and are unable to identify risk factors (Fante, 2019). A Pelvic Floor Health Knowledge Quiz was created by Al-Deges in order to evaluate the level of knowledge about pelvic floor and pelvic floor dysfunction in women and men in our country (Al-Deges, 2019).

In line with this information, the aim of our study is to determine the level of knowledge about pelvic floor and pelvic floor dysfunctions in women and men of different age groups. The target audience of our research is male and female individuals over the age of 18, and our research will be conducted online. As a result of the information we obtained from our research, the level of knowledge of individuals living in our country about pelvic floor and pelvic floor dysfunctions will be determined and the literature will be contributed. In addition, by determining the missing information of the society about the pelvic floor, contribution will be made to the development of appropriate intervention methods in order to eliminate the deficiencies in this area and to increase the level of awareness.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants over the age of 18
* Volunteering to participate in research

Exclusion Criteria:

* Not answering all questions in the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy people in Turkey
Sampling Method: Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Health Knowledge Quiz | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Berivan Beril Kiliç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008 May;27(3):379-87. doi: 10.1037/0278-6133.27.3.379. PMID 18624603
- [Background] AL-DEGES, W. (2019). Pelvik Taban Sağlığı Bilgi Testi Geliştirme, Geçerlik ve Güvenirliği (Doctoral dissertation, Ankara Yıldırım Beyazıt Üniversitesi Sağlık Bilimleri Enstitüsü).
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Arbuckle JL, Parden AM, Hoover K, Griffin RL, Richter HE. Prevalence and Awareness of Pelvic Floor Disorders in Female Adolescents Seeking Gynecologic Care. J Pediatr Adolesc Gynecol. 2019 Jun;32(3):288-292. doi: 10.1016/j.jpag.2018.11.010. Epub 2018 Dec 6. PMID 30529498
- [Background] Arnouk A, De E, Rehfuss A, Cappadocia C, Dickson S, Lian F. Physical, Complementary, and Alternative Medicine in the Treatment of Pelvic Floor Disorders. Curr Urol Rep. 2017 Jun;18(6):47. doi: 10.1007/s11934-017-0694-7. PMID 28585105
- [Background] Cardoso AMB, Lima CROP, Ferreira CWS. Prevalence of urinary incontinence in high-impact sports athletes and their association with knowledge, attitude and practice about this dysfunction. Eur J Sport Sci. 2018 Nov;18(10):1405-1412. doi: 10.1080/17461391.2018.1496146. Epub 2018 Jul 19. PMID 30025510
- [Background] Cohen D, Gonzalez J, Goldstein I. The Role of Pelvic Floor Muscles in Male Sexual Dysfunction and Pelvic Pain. Sex Med Rev. 2016 Jan;4(1):53-62. doi: 10.1016/j.sxmr.2015.10.001. Epub 2016 Jan 8. PMID 27872005
- [Background] Falvey L, Salameh F, O'Sullivan OE, O'Reilly BA. What Does Your Pelvic Floor Do for You? Knowledge of the Pelvic Floor in Female University Students: A Cross-sectional Study. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e457-e464. doi: 10.1097/SPV.0000000000000962. PMID 33109928
- [Background] Fante JF, Silva TD, Mateus-Vasconcelos ECL, Ferreira CHJ, Brito LGO. Do Women have Adequate Knowledge about Pelvic Floor Dysfunctions? A Systematic Review. Rev Bras Ginecol Obstet. 2019 Aug;41(8):508-519. doi: 10.1055/s-0039-1695002. Epub 2019 Aug 26. PMID 31450258
- [Background] Güngör M, Çetinkaya E. (2009). Pelvik taban yetmezliği, pelvik organ prolapsusu ve pelvik tabanı disfonksiyonları. Editör: Yalçın Ö. Temel Ürojinekoloji. İstanbul, Nobel Tıp Kitapevleri, s: 33-34.
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA) / International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016 Feb;27(2):165-94. doi: 10.1007/s00192-015-2932-1. PMID 26755051
- [Background] Hill AM, McPhail SM, Wilson JM, Berlach RG. Pregnant women's awareness, knowledge and beliefs about pelvic floor muscles: a cross-sectional survey. Int Urogynecol J. 2017 Oct;28(10):1557-1565. doi: 10.1007/s00192-017-3309-4. Epub 2017 Mar 14. PMID 28293791
- [Background] Kahyaoğlu Süt, H , Küçükkaya, B . (2018). Kadınların Pelvik Taban Kas Egzersizleri Bilgi ve Uygulama Durumları. Süleyman Demirel Üniversitesi Sağlık Bilimleri Dergisi, 9 (3) , 15-20 . DOI: 10.22312/sdusbed.411894.
- [Background] Lai HH, Hsu EI, Teh BS, Butler EB, Boone TB. 13 years of experience with artificial urinary sphincter implantation at Baylor College of Medicine. J Urol. 2007 Mar;177(3):1021-5. doi: 10.1016/j.juro.2006.10.062. PMID 17296403
- [Background] Lakhoo J, Khatri G, Elsayed RF, Chernyak V, Olpin J, Steiner A, Tammisetti VS, Sundaram KM, Arora SS. MRI of the Male Pelvic Floor. Radiographics. 2019 Nov-Dec;39(7):2003-2022. doi: 10.1148/rg.2019190064. PMID 31697623
- [Background] Liu J, Tan SQ, Han HC. Knowledge of pelvic floor disorder in pregnancy. Int Urogynecol J. 2019 Jun;30(6):991-1001. doi: 10.1007/s00192-019-03891-3. Epub 2019 Feb 19. PMID 30783706
- [Background] Machin SE, Mukhopadhyay S. Pelvic organ prolapse: review of the aetiology, presentation, diagnosis and management. Menopause Int. 2011 Dec;17(4):132-6. doi: 10.1258/mi.2011.011108. Epub 2011 Nov 25. PMID 22120945
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Neels H, Wyndaele JJ, Tjalma WA, De Wachter S, Wyndaele M, Vermandel A. Knowledge of the pelvic floor in nulliparous women. J Phys Ther Sci. 2016 May;28(5):1524-33. doi: 10.1589/jpts.28.1524. Epub 2016 May 31. PMID 27313364
- [Background] Parden AM, Griffin RL, Hoover K, Ellington DR, Gleason JL, Burgio KL, Richter HE. Prevalence, Awareness, and Understanding of Pelvic Floor Disorders in Adolescent and Young Women. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):346-54. doi: 10.1097/SPV.0000000000000287. PMID 27171318
- [Background] Sun C, Hull T, Ozuner G. Risk factors and clinical characteristics of rectal prolapse in young patients. J Visc Surg. 2014 Dec;151(6):425-9. doi: 10.1016/j.jviscsurg.2014.07.013. Epub 2014 Sep 18. PMID 25242503
- [Background] Verbeek M, Hayward L. Pelvic Floor Dysfunction And Its Effect On Quality Of Sexual Life. Sex Med Rev. 2019 Oct;7(4):559-564. doi: 10.1016/j.sxmr.2019.05.007. Epub 2019 Jul 24. PMID 31351916
- [Background] Wallace SL, Miller LD, Mishra K. Pelvic floor physical therapy in the treatment of pelvic floor dysfunction in women. Curr Opin Obstet Gynecol. 2019 Dec;31(6):485-493. doi: 10.1097/GCO.0000000000000584. PMID 31609735